CLINICAL TRIAL: NCT00004559
Title: Fatty Acid Antiarrhythmia Trial (FAAT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 127; R01HL062154 (NIH)
Record Dates: First submitted 2000-02-09; First posted 2000-02-10 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-11

CONDITIONS: Arrhythmia; Heart Diseases; Tachycardia, Ventricular; Ventricular Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Diseases; Tachycardia, Ventricular; Ventricular Fibrillation

INTERVENTIONS:
Behavioral: dietary polyunsaturated fatty acid

SUMMARY:
To determine if the dietary N-3 class of polyunsaturated fatty acids (PUFAs) provided in the diet largely from marine fish oils would prevent fatal ventricular tachycardia (VT) or ventricular fibrillation (VF).

DETAILED DESCRIPTION:
BACKGROUND:

Sudden death is a common manifestation of ischemic heart disease and therefore of great public health concern. Unfortunately several promising antiarrhythmic drugs proved not to be effective in preventing sudden deaths. This project would test whether a relatively inexpensive and presumably innocuous therapy, fish oil supplements, can prevent life-threatening arrhythmias. There is ample basic evidence that n-3 fatty acids contained in fish oil supplements may suppress arrhythmias, and a clinical trial seems warranted.

DESIGN NARRATIVE:

Prospective, randomized, placebo-controlled, double-blind. Patients were randomized to 4 grams per day of a PUFA fish oil supplement versus an olive oil placebo. The number of therapeutic discharges were recorded from the ICDs and then confirmed from the recorded electrocardiogram strips with the kinds of arrhythmias which had induced the ICD response. The primary end point, time to first ICD event for ventricular tachycardia or fibrillation (VT or VF) confirmed by stored electrograms or death from any cause, was analyzed by intention to treat.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Study Completion 2002-02 (Actual)

REFERENCES:
- [Background] Leaf A, Albert CM, Josephson M, Steinhaus D, Kluger J, Kang JX, Cox B, Zhang H, Schoenfeld D; Fatty Acid Antiarrhythmia Trial Investigators. Prevention of fatal arrhythmias in high-risk subjects by fish oil n-3 fatty acid intake. Circulation. 2005 Nov 1;112(18):2762-8. doi: 10.1161/CIRCULATIONAHA.105.549527. PMID 16267249